CLINICAL TRIAL: NCT03914703
Title: Post-market Clinical Follow-up Study to Collect Safety, Performance and Clinical Data of the EZPass Suture Passer (Instrumentation) and Precision Flexible Reamers (Instrumentation)- A Retrospective Consecutive Series Study
Brief Title: MDR EZ Pass and Precision Flexible Reamer
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-32SM
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Anterior Cruciate Ligament Injury; Rotator Cuff Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- EZ Pass Suture Passer: Patients who have surgery using the EZ Pass Suture Passer Instrument either in rotator cuff or soft tissue repair
  Interventions: Procedure: EZ Pass Suture Passer
- Precision Flexible Reamer: Patients who have surgery using the Precision Flexible Reamer Instrument in ACL repair
  Interventions: Procedure: EZ Pass Suture Passer

INTERVENTIONS:
Procedure: EZ Pass Suture Passer — Instruments used to help with rotator cuff or ACL repair

SUMMARY:
The objective of this study is to confirm the safety and performance on the EZPass Suture Passer Instrumentation and the Precision Flexible Reamer Instrumentation.

DETAILED DESCRIPTION:
The primary objective of the study is to assess performance, clinical benefits and safety of the EZPass Suture Passer and the Precision Flexible Reamer Instrumentation.

Performance and clinical benefits will be assessed through an operative survey conducted immediately following intraoperative surgery to determine if the device performed as expected.

Safety will be assessed by recording and analyzing the incidence and frequency of complications, adverse events, and intra-operative revisions.

ELIGIBILITY:
Inclusion Criteria

* EZ Pass Suture Passer:

  - Intended as an open or arthroscopic instrument utilized in conjunction with a nitinol wire or nylon monofilament to aid in passing suture through soft tissue.
* Precision Flexible Reamer:

  * This device is a hand held, or hand-manipulated device, intended to be used in ACL and PCL reconstruction surgeries and is intended for medical purposes to manipulate tissue, or for use with other devices in these surgeries.

Exclusion Criteria

* EZ Pass Suture Passer:

  - Any use other than the approved uses indicated in the Instructions for Use (IFU).
* Precision Flexible Reamer:

  * Any use other than the approved uses indicated in the Instructions for Use (IFU).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population should be a consecutive series of subjects where the EZPass Suture Passer or Precision Flexible Reamer instrumentation will be used.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Osborn, Study Director — Zimmer Biomet
Locations (1):
- OrthoCarolina, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- EZ Pass Suture Passer: Patients who have surgery using the EZ Pass Suture Passer Instrument either in rotator cuff or soft tissue repair
  EZ Pass Suture Passer: open or arthroscopic instrument utilized in conjunction with a nitinol wire or nylon monofilament to aid in passing suture through soft tissue
- Precision Flexible Reamer: Patients who have surgery using the Precision Flexible Reamer Instrument in ACL repair
  Precision Flexible Reamer: handheld/hand-manipulated device intended to be used in ACL or PCL reconstruction surgeries, intended to manipulate tissue or in conjunction with other devices
Period: Overall Study
Arm/Group | EZ Pass Suture Passer | Precision Flexible Reamer
Started | 51 | 22
Completed | 51 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients who have received either the EZ Pass Suture Passer or the Precision Flexible Reamer.
Groups:
- Total: Total of all reporting groups
Arm/Group | EZ Pass Suture Passer | Precision Flexible Reamer | Total
Number analyzed (Participants) | 51 | 22 | 73
Age, Continuous [Mean (Full Range); unit: years] | 54.1 [20.0 to 78.0] | 30.6 [18.0 to 54.0] | 47.02 [18.0 to 78.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 9 | 31
  Male | 29 | 13 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Performance of Instruments (EZ Pass Suture Passer and Precision Flexible Reamer)
Description: Questionnaire was completed to assess if the Instrument Performed as Expected. Surgeon provided yes/no answers on their opinion if the instrument performed as expected during the procedure.
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Groups:
- Precision Flexible Reamer: Patients who have surgery using the Precision Flexible Reamer Instrument in ACL repair
  Precision Flexible Reamer: A handheld device intended to be used in ACL and PCL reconstruction surgeries to manipulate tissue, or in conjunction with other devices in these surgeries.
Arm/Group | EZ Pass Suture Passer | Precision Flexible Reamer
Number analyzed (Participants) | 51 | 22
Participants
  Performed as Expected | 49 | 22
  Did Not Perform as Expected | 2 | 0

2. Primary Outcome: Absence of Instrument Related Serious Adverse Events
Description: This outcome will measure the frequency of instrument related serious adverse events
Time Frame: Intraoperative
Population: Questionnaire will be used to assess whether subjects had any instrument-related serious adverse events. Responses are yes/no.
Measure: Count of Participants; unit: Participants
Arm/Group | EZ Pass Suture Passer | Precision Flexible Reamer
Number analyzed (Participants) | 51 | 22
Participants
  Subject with No Instrument-Related Serious Adverse Event | 51 | 22
  Subject with Instrument-Related Serious Adverse Event | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events occurring on the day of surgery were reported and assessed.
Groups:
- Precision Flexible Reamer: Patients who have surgery using the Precision Flexible Reamer Instrument in ACL repair
  Precision Flexible Reamer: handheld device intended to be used in ACL and PCL reconstruction surgeries to manipulate tissue, or in conjunction with other devices in these surgeries.
Arm/Group | EZ Pass Suture Passer | Precision Flexible Reamer
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/22
Other Adverse Events (participants affected / at risk) | 5/51 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EZ Pass Suture Passer (N=51) | Precision Flexible Reamer (N=22)
Instrument Malfunction (Surgical and medical procedures) | 2 | 2 — Kite broke when grabbed with Suture Grasper
Instrument Malfunction (Surgical and medical procedures) | 3 | 0 — Kite would not advance

LIMITATIONS AND CAVEATS:
Among the limitations of the study was that it was comprised of a single center of non-randomized enrollment. Additional limitations include no patient reported outcome measures or post-operative follow-up visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT03914703/Prot_SAP_000.pdf